CLINICAL TRIAL: NCT02465801
Title: Efficacy and Safety Phase II Study of Recombinant Human Serum Albumin/Granulocyte Colony-Stimulating Factor Fusion Protein for Injection to Prevent Neutrophilic Granulocytopenia Among Chemotherapy Patients
Brief Title: Study of Recombinant Human Serum Albumin/Granulocyte Colony-Stimulating Factor Fusion Protein
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin SinoBiotech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RG01N-0778
Record Dates: First submitted 2014-11-17; First posted 2015-06-08 (Estimated); Last update posted 2017-07-18 (Actual); Status verified 2014-11

CONDITIONS: Chemotherapy-induced Neutropenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Experimental): Intervention: HSA-GCSF 1.2 mg
  Drug: TE or TEC TE: Taxotere+Epirubicin Taxotere (75mg/m2) and Epirubicin (75mg/m2), IV on day 1 of each 21 chemotherapy cycle.
  TEC:Taxotere+Epirubicin+Cyclophosphamide Taxotere (75mg/m2),Epirubicin (75mg/m2) and Cyclophosphamide (500mg/m2), IV on day 1 of each 21 chemotherapy cycle.
  Recombinant Human Serum Albumin/Granulocyte Colony-Stimulating Factor Fusion Protein（1.2mg）will be injected subcutaneously at night o'clock a.m. in the 3rd and 7th day of per chemotherapy cycle. After the injection, stop administrating if Absolute Neutrophil Count (ANC) in peripheral blood exceeded 1.5×109/L at two contiguous times at least. If not up to standard, investigator should decide whether or not the third administration.
  Interventions: Drug: HSA-GCSF 1.2 mg
- Group 2 (Experimental): Intervention:HSA-GCSF 1.5 mg
  Drug: TE or TEC TE: Taxotere+Epirubicin Taxotere (75mg/m2) and Epirubicin (75mg/m2), IV on day 1 of each 21 chemotherapy cycle.
  TEC:Taxotere+Epirubicin+Cyclophosphamide Taxotere (75mg/m2),Epirubicin (75mg/m2) and Cyclophosphamide (500mg/m2), IV on day 1 of each 21 chemotherapy cycle.
  Recombinant Human Serum Albumin/Granulocyte Colony-Stimulating Factor Fusion Protein（1.5mg）will be injected subcutaneously at night o'clock a.m. in the 3rd and 7th day of per chemotherapy cycle. After the injection, stop administrating if Absolute Neutrophil Count (ANC) in peripheral blood exceeded 1.5×109/L at two contiguous times at least. If not up to standard, investigator should decide whether or not the third administration.
  Intervention: Drug: TE or TEC
  Interventions: Drug: HSA-GCSF 1.5 mg
- Group 3 (Active Comparator): Intervention: GCSF
  Drug: TE or TEC TE: Taxotere+Epirubicin Taxotere (75mg/m2) and Epirubicin (75mg/m2), IV on day 1 of each 21 chemotherapy cycle.
  TEC:Taxotere+Epirubicin+Cyclophosphamide Taxotere (75mg/m2),Epirubicin (75mg/m2) and Cyclophosphamide (500mg/m2), IV on day 1 of each 21 chemotherapy cycle.
  Recombinant Human Granulocyte Colony-Stimulating Factor Injection (5μg/kg/day) will be injected subcutaneously at night o'clock a.m. from the 3rd of per chemotherapy cycle. After the injection, stop administrating if Absolute Neutrophil Count (ANC) in peripheral blood exceeded 1.5×109/L at two contiguous times at least. The maximum of usage was continuous 14 days.
  Intervention: Drug: TE or TEC
  Interventions: Drug: GCSF

INTERVENTIONS:
Drug: HSA-GCSF 1.2 mg — Human Serum Albumin GCSF 1.2mg at day 3 and Day 7
  Arms: Group 1
Drug: HSA-GCSF 1.5 mg — Human Serum Albumin GCSF 1.5 mg at day 3 and Day 7
  Arms: Group 2
Drug: GCSF — GCSF 5 mcg/kg/day
  Arms: Group 3

SUMMARY:
The purpose of this study is to evaluate the dosages of recombinant human serum albumin/granulocyte colony-stimulating factor fusion protein by injection for preventing neutrophilic granulocytopenia among chemotherapy patients.

Conduct Pharmacokinetics (PK) study on recombinant human serum albumin/granulocyte colony-stimulating factor fusion protein with recombinant human granulocyte colony-stimulating factor injection as a control.

DETAILED DESCRIPTION:
* Brief Protocol: Treat the patients taking Taxotere+Epirubicin+Cyclophosphamide (TEC) treatment or Taxotere+Epirubicin (TE) treatment chemotherapy with the study medicine or positive control during the period between two chemotherapy treatments.
* Positive control：recombinant human granulocyte colony-stimulating factor injection.
* Targeted patients: breast cancer
* Grouping: Group 1: 1.2 mg recombinant human serum albumin/granulocyte colony-stimulating factor fusion protein with TEC or TE treatment; Group 2: 1.5 mg recombinant human serum albumin/granulocyte colony-stimulating factor fusion protein with TEC or TE treatment; Group 3: positive control with TEC or TE treatment.
* Number of patients: 216
* Concomitant medicines will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65.
* Diagnosed breast cancer, suitable for TEC or TE .
* ECOG performance status 0 or 1.
* Adjuvant chemotherapy; new adjuvant chemotherapy; newly diagnosed class Ⅳ and prior chemotherapy.
* ANC≥1.5×10 9/L, PLT≥100×10 9/L. No bone marrow metastasis,blood coagulation function normally, no Hemorrhagic tendency.
* No obvious abnormal ecg examination.
* TBIL, ALT, AST≤2.5×ULN (≤5×ULN if presence of hepatic metastases).
* Cr, BUN≤2.5×ULN.
* Signed informed consent.

Exclusion Criteria:

* Chemotherapy within past 4 weeks
* Uncontrolled inflammatory disease,axillary temperature≥38℃.
* Merging other malignant tumor
* Pregnancy or nursing status.
* Participation in another clinical trial with and investigational product within 3 months prior to study entry.
* Severe diabetes mellitus, or poor blood sugar controller.
* Allergic disease or allergic constitution. History of protein allergy.
* History of drug addiction and alcoholism.
* Hematopoietic stem cell transplantation or organ transplantation.
* Chronic disease of severe cardiac, kidney and liver.
* Other conditions that would be excluded from this study according to doctors'judgment

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2014-12-16 (Actual); Primary Completion 2015-12-23 (Actual); Study Completion 2016-04-26 (Actual)

PRIMARY OUTCOMES:
The mean of duration for class IV neutrophilic granulocytopenia | 4 weeks

SECONDARY OUTCOMES:
The mean of duration for class IV neutrophilic granulocytopenia | 8 weeks
The mean of duration for ANC up to 2.0×109/L | 8 weeks
ANC | 8 weeks
The usage of antibiotics | 8 weeks
febrile neutropenia | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Binhe Xu, MD, Principal Investigator — CAMS
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Scienses, Beijing, China

REFERENCES:
- [Derived] Chen S, Han Y, Ouyang Q, Lu J, Zhang Q, Yang S, Wang J, Huang H, Liu H, Shao Z, Li H, Chen Z, Sun S, Geng C, Lu J, Sun J, Wang J, Xu B. Randomized and dose-escalation trials of recombinant human serum albumin /granulocyte colony-stimulating factor in patients with breast cancer receiving anthracycline-containing chemotherapy. BMC Cancer. 2021 Mar 31;21(1):341. doi: 10.1186/s12885-021-08093-z. PMID 33789616